CLINICAL TRIAL: NCT02664389
Title: Targeted Next-generation Sequencing Panel for Identification of Germline Mutations in Early Onset Cancers With Sporadic or Hereditary Presentation
Acronym: PANEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/160/HP
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Ovarian Cancer; Colorectal Cancer; Pediatric Cancers; Multiple Primary Malignant Tumours
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Genetic analysis of patient with early-onset breast cancer (Experimental): Sequencing of 200 selected genes in patient with early-onset breast cancer without genomic alterations of BRCA1, BRCA2 or TP53
  Interventions: Genetic: Genetic analysis
- Genetic analysis of patient with early-onset ovarian cancer (Experimental): Sequencing of 200 selected genes in patient with early-onset ovarian cancer without genomic alterations of BRCA1, BRCA2
  Interventions: Genetic: Genetic analysis
- Genetic analysis of patient with pediatric cancer (Experimental): Sequencing of 200 selected genes in patient with pediatric cancer without genomic alteration of TP53
  Interventions: Genetic: Genetic analysis
- Genetic analysis of patient with early-onset colorectal cancer (Experimental): Sequencing of 200 selected genes in patient with early-onset colorectal cancer without genomic alteration of APC, MUTYH, SMAD4, BMPR1A, PTEN or STK11 in case of adenomatous polyposis or hamartoma presentation or without genomic alteration of MSH2, MLH1 or MSH6 in case of HNPCC presentation
  Interventions: Genetic: Genetic analysis
- Genetic analysis of patient with multiple primary tumors (Experimental): Sequencing of 200 selected genes in patient with Multiple primary malignant tumors without syndromic presentation
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis — Sequencing of 200 selected genes in the different study populations

SUMMARY:
Despite relevant clinical and/or familial presentations suggesting a hereditary predisposition (early-onset, multiple primary tumors, familial aggregation), targeted genomic analysis based on the phenotype are often non contributive. As somatic cancer genes are limited, the hypothesis is that the targeted next-generation sequencing of 200 genes, selected for their implications in cancers may contribute to the understanding of many selected patients' presentation by the identification of germline deleterious mutations, and may identified phenotype overlapping and/or mosaicisms. The focus will be put on early-onset breast, ovarian, colorectal cancer or pediatric cancers and multiple primary tumors.

ELIGIBILITY:
Inclusion Criteria :

* Older than 18 or parental agreement in case of children.

For patient with early-onset breast cancer :

* Invasive breast cancer, regardless of histological type or stage, diagnosed before 31 years.
* Sporadic or familial presentation
* No genomic alterations of BRCA1, BRCA2 or TP53

For patient with early-onset ovarian cancer :

* Invasive ovarian cancer, regardless of histological type or stage, diagnosed before 41 years.
* Sporadic or familial presentation
* No genomic alterations of BRCA1, BRCA2

Patient with early-onset colorectal cancer :

* Invasive colorectal cancer diagnosed before 31 years.
* Sporadic or familial presentation
* No genomic alteration of MSH2, MLH1 or MSH6 in case of HNPCC presentation
* No genomic alteration of APC, MUTYH, SMAD4, BMPR1A, PTEN or STK11 in case of adenomatous polyposis or hamartoma presentation

Patient with pediatric cancer :

* Non haematological tumour diagnosed before 16 years, with Li-Fraumeni presentation.
* No genomic alteration of TP53

Patient with Multiple primary malignant tumours :

* Multiple synchronous or metachronous primary malignant tumors with early-onset
* No syndromic presentation

Exclusion Criteria:

* Any already known deleterious mutations according to the patient's phenotype

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Frequency of germline deleterious mutations | Day 1
  Frequency of germline deleterious mutations will be assessed for the 200 selected genes using next generation sequencing method

CONTACTS AND LOCATIONS:
Overall Officials: Thierry FREBOURG, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No